CLINICAL TRIAL: NCT02368626
Title: Evaluation of the Safety and Efficacy of the EndyMed Pro™ System Using Radiofrequency (RF) Micro-needles Fractional Skin Remodeling Handpiece (Intensif) for Wrinkle Reduction and Lifting - a Post Marketing Study
Brief Title: Safety and Efficacy of the EndyMed Pro System Using RF Micro-needles Fractional Skin Remodeling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: EndyMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-FR-01
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RF ablation treatment (Experimental): 'EndyMed Pro™ RF Micro-Needles' - RF ablation treatments for wrinkle appearance reduction
  Interventions: Device: EndyMed Pro™ RF Micro-Needles

INTERVENTIONS:
Device: EndyMed Pro™ RF Micro-Needles — RF Micro-needles ablation treatments

SUMMARY:
The need for cosmetic facial enhancement procedures with minimal down time and low risk has led to the development of methods for non-surgical skin rejuvenation. Various ablative lasers were developed, which remove the full skin surface in a controlled manner. However, the prolonged recovery and the significant risks prompted the development of fractional lasers which ablate the skin in a fractional manner, leaving untreated areas to improve healing process. In the past few years, fractional RF systems have been introduced that enable controlled skin resurfacing accompanied with dermal collagen remodeling. System using focused ultrasound , coagulating small volume of tissue in the dermis , have shown a lifting effect.8 Similar to these devices the EndyMed Pro™ System with RF Micro-Needles handpiece (INTENSIF) enables fractional skin coagulation with dermal heating for the reduction of wrinkles together with a lifting effect.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients age 35-60 with facial condition as required by the treatment.
* Subjects with Fitzpatrick elasticity level of 4 and above
* Subject able to comprehend and sign informed consent for participation in this study.
* Subject must commit to all treatments and follow-up visits.
* Subjects must approve the use of their B&A photos by the doctor and EndyMed

Exclusion Criteria:

* Subjects with implanted pacemakers, arrhythmias or any other electronic implanted device or severe known heart disorder
* Subjects with any implantable metal device in the treatment area.
* Subjects on any medication that would affect the characteristic of the skin (medical or hormonal), such as "Accutane", within the past 3 months.
* Subjects that have had any other invasive or noninvasive method of skin therapy hair removal, filers or Botox, performed in the past 3 months (in the treated area).
* Subjects who are scheduled or planned for any other invasive or noninvasive method of skin therapy in the treatment area at the period of the study.
* Subjects who have any form of suspicious lesion on the treatment area.
* Subjects with hypertrophic scarring, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Pregnant or lactating Subjects.
* Subjects with Epilepsy or severe migraines.
* Subjects with permanent makeup/ tattoo/ body piercing (in the treated area).
* Subjects with any Infection / abscess / pains in treatment target area.
* History of any kind of cancer
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regime.
* Any surgical procedure in the treatment area within the last 3 months or before complete healing.
* Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.
* Treating over the thyroid, breast or any other sensitive area.
* Subjects who suffer from autoimmune disorders or diabetes.
* Subjects using blood thinning medications.
* Subjects with clotting disorders.
* Subjects on drugs or psychologically determined unsuitable for the study.
* Subject is suffering extreme general weakness.
* Subject objects to the study protocol or unwilling to sign a consent form. Concurrent participation in any other clinical study.
* Any other condition that exclude the patient from the evaluation according to the physician judgment.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of the EndyMed ProTM Intensif handpiece for wrinkle reduction and lifting, measured by Adverse events occurrence | 5 months
  Adverse events occurrence

SECONDARY OUTCOMES:
To evaluate the efficacy of the EndyMed ProTM Intensif handpiece for wrinkle reduction and lifting, measured by wrinkle appearance reduction | 5 months
  wrinkle appearance reduction

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, Dr, Principal Investigator — Tennessee Clinical Research Center, Nashville, Tennessee, USA; Mark Taylor, Dr, Principal Investigator — Gateway Aesthetic Institute and Laser Center, Salt Lake City, Utah, USA; Kenneth Rothaus, Dr, Principal Investigator — Ageless Plastic Surgery, New York, NY, USA; Yohei Tanaka, Dr, Principal Investigator — Clinica Tanaka Plastic and Reconstructive Surgery and Anti-aging Center, Tokyo, Japan